CLINICAL TRIAL: NCT02908321
Title: Cognitive Behavioural Therapy for Anxiety Disorder in Children With Co-morbid Autism Spectrum Disorder
Brief Title: CBT for Anxiety Disorder in Children With Co-morbid ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-2018
Record Dates: First submitted 2016-09-07; First posted 2016-09-20 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2019-04

CONDITIONS: Randomized Treatment Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Active Comparator)
  Interventions: Behavioral: CBT
- WL (No Intervention)

INTERVENTIONS:
Behavioral: CBT — The group based manualised CBT intervention consists of The Cool Kids Anxiety Program: Autism Spectrum Disorder Adaptation (Cool Kids ASD).
  Other Names: Cool Kids ASD
  Arms: CBT

SUMMARY:
Children with Autism Spectrum Disorder (ASD) often have other difficulties as a result of the disorder. Up to half of the children with ASD are thought to suffer with anxiety in a way that interferes with their wellbeing and every day functioning. In this project the investigators will study the effect of the group program The Cool Kids Anxiety Program: Autism Spectrum Disorder Adaptation (Cool Kids ASD) - an anxiety treatment program specific developed for children with ASD. The investigators expect a decrease in the overall anxiety level together with an increase in the ability of handling anxiety.

DETAILED DESCRIPTION:
The primary objective is to investigate the effect of a manualised Cognitive Behavioural Therapy (CBT) programme The Cool Kids Anxiety Program: Autism Spectrum Disorder Adaptation (Cool Kids ASD) for anxiety disorder adapted to children with Autism Spectrum Disorder (ASD) in a waitlist controlled design.

The investigators will investigate treatment effects on anxiety diagnosis and anxiety symptoms. Further, the investigators will investigate outcomes related to general functioning, co-morbid psychiatric disorders (Obsessive-Compulsive Disorder (OCD), hyperkinetic disorder and depression) and level of ASD symptoms (social and communicative skills).

ELIGIBILITY:
Inclusion Criteria:

* ASD
* Anxiety (not necessary diagnosed)

Exclusion Criteria:

* IQ under 70
* Not meeting diagnostic criteria for primary anxiety diagnosis on ADIS
* Active psychosis
* Untreated ADHD
* Families not able to follow program

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2016-08; Primary Completion 2019-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule for DSM-IV: Parent & Child interview schedule (ADIS/CP). | Change from baseline interview results at 14 weeks
  ADIS/CP is a structured interview involving both child and parents designed to assess for current episodes of anxiety disorders, and to permit differential diagnosis among the anxiety disorders according to DSM-IV criteria.
Anxiety Disorders Interview Schedule for DSM-IV: Parent & Child interview schedule (ADIS/CP). | Change from baseline interview results at 3 months
  ADIS/CP is a structured interview involving both child and parents designed to assess for current episodes of anxiety disorders, and to permit differential diagnosis among the anxiety disorders according to DSM-IV criteria.

SECONDARY OUTCOMES:
Spence Children's Anxiety Scale (SCAS), | Change from baseline results at 14 weeks
  SCAS is a questionnaire for children and parents assessing the severity of anxiety symptoms broadly in line with the dimensions of anxiety disorder proposed by the DSM-IV. The scale assesses six domains of anxiety including generalized anxiety, panic/agoraphobia, social phobia, separation anxiety, obsessive-compulsive disorder and physical injury fears.
Spence Children's Anxiety Scale (SCAS), | Change from baseline results at 3 months
  SCAS is a questionnaire for children and parents assessing the severity of anxiety symptoms broadly in line with the dimensions of anxiety disorder proposed by the DSM-IV. The scale assesses six domains of anxiety including generalized anxiety, panic/agoraphobia, social phobia, separation anxiety, obsessive-compulsive disorder and physical injury fears.
Children's Anxiety Life Inference Scale (CALIS) | Change from baseline results at 14 weeks
  CALIS is designed to assess life interference attributed to fears and worries from child and parent perspectives. The measure targets interference on the child's life and on the parent's/family's life.
Children's Anxiety Life Inference Scale (CALIS) | Change from baseline results at 3 months
  CALIS is designed to assess life interference attributed to fears and worries from child and parent perspectives. The measure targets interference on the child's life and on the parent's/family's life.
Children's Automatic Thoughts Scale (CATS). | Change from baseline results at 14 weeks
  CATS is a developmentally sensitive, general measure of negative self-statements across both internalizing and externalizing problems. Four separate subscales of cognitive content are assessed including physical threat, social threat, personal failure, and hostility.
Children's Automatic Thoughts Scale (CATS). | Change from baseline results at 3 months
  CATS is a developmentally sensitive, general measure of negative self-statements across both internalizing and externalizing problems. Four separate subscales of cognitive content are assessed including physical threat, social threat, personal failure, and hostility.

OTHER OUTCOMES:
Attention Deficit/Hyperactive Disorder-Rating Scale (ADHD-RS) | Change from baseline results at 14 weeks
Attention Deficit/Hyperactive Disorder-Rating Scale (ADHD-RS) | Change from baseline results at 3 months
Social Responsiveness Scale (SRS) | Change from baseline results at 14 weeks
Social Responsiveness Scale (SRS) | Change from baseline results at 3 months
Strength and Difficulties Questionnaire (SDQ) | Change from baseline results at 14 weeks
Strength and Difficulties Questionnaire (SDQ) | Change from baseline results at 3 months
The WHO-five Well-being Index (WHO-5) | Change from baseline results at 14 weeks
The WHO-five Well-being Index (WHO-5) | Change from baseline results at 3 months
Adaptive Behaviour Assessment System, Second Edition (ABAS-II) | Change from baseline results at 14 weeks
Adaptive Behaviour Assessment System, Second Edition (ABAS-II) | Change from baseline results at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Child and Adolescent Psychiatry, Risskov, Region of Midtjylland, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be on group basis only

REFERENCES:
- [Derived] Kilburn TR, Sorensen MJ, Thastum M, Rapee RM, Rask CU, Arendt KB, Thomsen PH. Rationale and design for cognitive behavioral therapy for anxiety disorders in children with autism spectrum disorder: a study protocol of a randomized controlled trial. Trials. 2018 Apr 2;19(1):210. doi: 10.1186/s13063-018-2591-x. PMID 29609630